CLINICAL TRIAL: NCT03578432
Title: Clinical Evaluation of Everolimus (a Rapamycin Analog) in Restoring Salivary Gland Function to Patients Treated With Radiotherapy for Head and Neck Cancer
Brief Title: Everolimus in Restoring Salivary Gland Function in Participants With Locally Advanced Head and Neck Cancer Treated With Radiation Therapy
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: UACC-PHX is no longer able to support the study and Novartis is unable to provide drug beyond December 2019.
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PHXB-17-0072-70-15; NCI-2018-00492 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CRAD001XUA274T; PHXB-17-0072-70-15 (Other: The University of Arizona Cancer Center); P30CA023074 (NIH)
Record Dates: First submitted 2018-06-15; First posted 2018-07-06 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Salivary Gland Dysfunction; Xerostomia; Head and Neck Cancer
Keywords: Xerostomia; Dry Mouth; Salivary Gland Dysfunction; Head and Neck Cancer; Mouth Cancer; Everolimus; Rapamycin; Neck Cancer; Saliva
MeSH Terms: conditions — Xerostomia; Head and Neck Neoplasms; Mouth Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive care (everolimus, saliva output testing) (Experimental): Participants receive everolimus PO QD for 5 days beginning 2 weeks after radiation treatment. Participants also undergo saliva output testing at baseline prior to radiation or chemoradiation treatment, after 3 weeks of RT/chemoRT, after 6 weeks of RT/chemoRT, prior to everolimus administration, at completion of the 5 day everolimus course, and at 1, 3, and 6 months after the completion of radiation or chemoradiation therapy.
  Interventions: Drug: Everolimus; Other: Laboratory Biomarker Analysis; Other: Survey Administration

INTERVENTIONS:
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001; Votubia; Zortress
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This early phase 1 trial studies the use of everolimus in restoring salivary gland function in participants with locally advanced head and neck cancer after concurrent chemoradiation or radiation therapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe the recovery of salivary gland function after administration of a 5-day course of everolimus, administered two weeks after completion of radiation or chemoradiation therapy.

SECONDARY OBJECTIVES:

I. To describe the decrease of saliva flow rates during radiation or chemoradiation therapy.

II. To describe the changes in saliva protein composition during radiation or chemoradiation therapy and following administration of a 5-day course of everolimus.

OUTLINE: This is an early phase 1 proof of principal study.

Participants receive everolimus orally (PO) once daily (QD) for 5 days beginning 2 weeks after completion of radiation or chemoradiation treatment. Participants also undergo saliva output testing at baseline prior to radiation or chemoradiation treatment, after 3 weeks of RT/chemoRT, after 6 weeks of RT/chemoRT, prior to everolimus administration, at completion of the 5 day everolimus course, and at 1, 3, and 6 months after the completion of radiation or chemoradiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Performance status Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
* Platelets ≥ 100 x 10^9/L
* Hemoglobin (Hgb) > 9 g/dL
* Total serum bilirubin ≤ 2.0 mg/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x upper limits of normal (ULN) (≤ 5 x ULN in patients with liver metastases)
* International normalized ratio (INR) ≤ 2
* Serum creatinine ≤ 1.5 x ULN
* Fasting serum cholesterol ≤ 300 mg/dL or ≤ 7.75 mmol/L and fasting triglycerides ≤ 2.5 x ULN

  * NOTE: in case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication
* Signed informed consent obtained prior to any screening procedures
* Patients with locally advanced squamous cell carcinoma of the head and neck, treated with curative intent either in the post-operative or definitive setting with high dose radiotherapy (≥ 50 Gy) with or without chemotherapy

Exclusion Criteria:

* Patients currently receiving anticancer therapies or who have received anticancer therapies within 2 weeks of the start of everolimus (including chemotherapy, radiation therapy, antibody based therapy, etc.)
* Known intolerance or hypersensitivity to everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus)
* Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral everolimus
* Uncontrolled diabetes mellitus as defined by glycated hemoglobin (HbA1c) > 8% despite adequate therapy; patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary
* Patients who have any severe and/or uncontrolled medical conditions such as:

  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤ 6 months prior to start of everolimus, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease
  * Symptomatic congestive heart failure of New York heart Association class III or IV
  * Active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and active and chronic hepatitis (i.e. quantifiable hepatitis B virus [HBV]-deoxyribonucleic acid [DNA] and/or positive hepatitis B virus surface antigen [HbsAg], quantifiable hepatitis C virus [HCV]-ribonucleic acid [RNA])
  * Known severely impaired lung function (spirometry and carbon monoxide diffusing capacity [DLCO] 50% or less of normal and oxygen [O2] saturation 88% or less at rest on room air)
  * Active, bleeding diathesis
* Chronic treatment with corticosteroids or other immunosuppressive agents; topical or inhaled corticosteroids are allowed
* Known history of human immunodeficiency virus (HIV) seropositivity
* Patients who have received live attenuated vaccines within 1 week of start of everolimus and during the study; patient should also avoid close contact with others who have received live attenuated vaccines; examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, Bacillus Calmette-Guerin (BCG), yellow fever, varicella and TY21a typhoid vaccines
* Patients who have a history of another primary malignancy, with the exceptions of: nonmelanoma skin cancer, and carcinoma in situ of the cervix, uteri, or breast from which the patient has been disease free for ≥ 3 years
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study
* Patients who are currently part of or have participated in any clinical investigation with an investigational drug within 1 month prior to dosing
* Pregnant or nursing (lactating) women
* Women of child-bearing potential (WOCBP) (including female pediatric patients who are menarcheal or who become menarcheal during the treatment), defined as all women physiologically capable of becoming pregnant, must use highly effective methods of contraception during the study and 8 weeks after; women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms); highly effective contraception methods include combination of any two of the following:

  * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example, hormone vaginal ring or transdermal hormone contraception; in case of use of oral contraception women should have been stable on the oral agent for a minimum of 3 months before taking everolimus
  * Total abstinence
  * Male partner sterilization; (the vasectomized male partner should be the sole partner for that subject)
  * Female sterilization have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks prior torandomization; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential
* Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Percent recovery of salivary gland function | At 3 months after completion of radiation or chemoradiation therapy
  The primary end point of the analysis will be the percent recovery of salivary gland function, with pre-everolimus treatment saliva flow rate as the denominator and the saliva flow rate at 3 months after completion of radiation or chemoradiation therapy as the numerator.

SECONDARY OUTCOMES:
Change of saliva flow rates | Up to 6 months after completion of radiation or chemoradiation therapy
  This will be measured during radiotherapy treatment at 3, 6 weeks, and prior to everolimus administration and the subsequent recovery of saliva flow rates at completion of the 5 day everolimus course and 1, 3 and 6 months after radiation therapy/chemoradiation therapy completion to determine the kinetics and stability of saliva flow rate recovery. Will be explored using graphical methods.
Saliva protein composition | Up to 6 months after completion of radiation or chemoradiation therapy
  Protein composition within the saliva will be measured and will be expressed as percent decrease and recovery of amylase at all available time points. Will be explored using graphical methods.
Total score obtained on Xerostomia Visual Analog Scale survey | Up to 6 months after completion of radiation or chemoradiation therapy
  Will be explored using graphical methods. Subjective assessment of salivary dysfunction. • Scale ranges: not difficult at all - very difficult. • Not difficult at all is considered better, very difficult is considered worse. Subscales are summed. Scale ranges: 1-5 = • 1 (Never), 2 (hardly ever), 3 (occasionally), 4 (fairly often), 5 (very often). • Sub scales are summed.
Total score obtained on Xerostomia Inventory Survey | Up to 6 months after completion of radiation or chemoradiation therapy
  Will be explored using graphical methods. Measures xerostomia symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Panayiotis Savvides, Principal Investigator — The University of Arizona Cancer Center at Dignity Health St. Joseph's Hospital and Medical Center
Locations (1):
- The University of Arizona Cancer Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT03578432/Prot_000.pdf